CLINICAL TRIAL: NCT02818556
Title: A Clinical Study Comparing Restylane® Silk and Belotero Balance® for the Treatment of Superficial, Vertical Perioral Lines
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Maas Clinic (Other)
Responsible Party: Principal Investigator, Corey S. Maas, M.D., Principal Investigator, The Maas Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RSB-2015
Record Dates: First submitted 2016-06-03; First posted 2016-06-29 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-06

CONDITIONS: Perioral Rhytids
MeSH Terms: interventions — belotero balance

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Restylane Right, Belotero Left (Other): Patients will receive one treatment with Restylane® Silk (right side of the face) and one treatment of Belotero Balance® (left side)
  Interventions: Drug: Restalyne Silk; Drug: Belotero Balance
- Restylane Left, Belotero Right (Other): Patients will receive one treatment with Restylane® Silk (left side of the face) and one treatment of Belotero Balance® (right side)
  Interventions: Drug: Restalyne Silk; Drug: Belotero Balance

INTERVENTIONS:
Drug: Restalyne Silk
Drug: Belotero Balance

SUMMARY:
This will be a single-center, randomized, evaluator-blinded, split-face clinical study design. Fifty patients will receive one treatment session consisting of Restylane® Silk (right side of the face) and Belotero Balance® (left side), or vice versa (1:1 dose conversion ratio) injections to the superficial, vertical perioral lines. Injections will be performed at the baseline visit. To ensure subject and investigator blinding, syringes will be prepared and labeled "1" and "2" immediately before subject attendance for injection by the sub-investigator. The same injection sites and techniques will be used on both sides of the face. Then, patients will follow-up on post-treatment day 7, 14, 30, 60, 90, 120, 150, 180.

ELIGIBILITY:
Inclusion Criteria:

* Patients exhibiting moderate [2] to severe [3] superficial, vertical perioral lines on the 5-point Merz® validated scale for assessment of superficial perioral lines
* Females and males in good general health over the age of 18 years old

Must be willing to give and sign a HIPAA form, informed consent form and a photographic release form

* Patient is planning to undergo Restylane® Silk and Belotero Balance® injections
* For female patient of childbearing potential, must have had a regular menstrual cycle prior to study entry (a female is considered of childbearing potential unless she is postmenopausal, without a uterus and/or both ovaries, or has had a bilateral tubal ligation) and is willing to use an acceptable form of birth control during the entire course of the study [i.e., acceptable methods of birth control are oral contraceptives, contraceptive patches/rings/implants Norplanit®, Depo-Provena®, double-barrier methods (e.g. condoms and spermicide), abstinence and vasectomies of partner with a documented second acceptable method of birth control should the patient become sexually active]. All systemic birth control measures must be in consistent use at least 30 days prior to study participation
* Negative urine pregnancy test results at the time of study entry (if applicable)
* Must be willing to comply with study regimen and complete the entire course of the study.

Exclusion Criteria:

* A patient with any uncontrolled systemic disease. A potential patient in whom therapy for a systemic disease is not yet stabilized will not be considered for entry into the study

A patient with a significant history or current evidence of a medical, psychological or other disorder that, in the investigator's opinion, would preclude enrollment into the study.

* A patient with a known hypersensitivity to any of the components of the study medications
* A patient who is actively smoking or plans to smoke at any time of the duration of this study
* A patient with an active skin condition/disease that might interfere with the diagnosis or evaluation of study parameters (i.e., atopic dermatitis, eczema, psoriasis, seborrheic dermatitis, herpes labialis)
* A patient planning any other cosmetic procedure to their facial area during the study period, other than the treatments that will be performed by the investigator
* A patient using any topical (prescription or over the counter) medicated creams, lotions, gels, balms, powders, etc. on the treatment areas during the study period
* A patient receiving any topical products containing alpha-hydroxy acids, salicylic acid, and vitamins C or D (includes derivatives thereof) on the perioral areas within 7 days prior to or during the study period, other than the study products
* A patient receiving any investigational drug and/or has had a microdermabrasion (light or medium skin peel) treatment on their perioral areas within 30 days prior to or during the study period
* A patient using any topical tretinoin product or derivative on their perioral areas within 12 weeks prior to or during the study period
* A patient receiving a chemical peel, any systemic steroids, a non-ablative laser, light or radio frequency treatment and/or has had a dermabrasion (deep skin peel) or ablative laser treatments on their perioral areas must have discontinued the drug/treatment and/or had the procedure at least 6 months prior to entering the study
* A patient that has previously been treated with botulinum toxin in the perioral areas within the past six months
* A patient that has previously been treated with dermal filler in the perioral areas within the past year
* A patient that with a history of allergic reaction to a dermal filler or lidocaine
* A patient that with a history of a permanent filler to the perioral areas
* A female patient who is pregnant, nursing an infant or planning a pregnancy during the study [throughout the course of the study, women of child-bearing potential must use reliable forms of contraception (i.e., oral contraceptive, intrauterine device, abstinence, or spermicides and condoms used in combination)]
* Current participation or participation within 30 days prior to the start of this study in a drug or other investigational research study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Change in Response to therapy as evaluated by investigator using 5-point Merz® Scale | Day 0, 7, 14, 30, 60, 90, 120, 150, 180
  Response to therapy on each side of the lip on day 0 (initial treatment), and subsequent post-treatment days 7, 14, 30, 60, 90, 120, 150, 180, as measured by the blinded evaluator: A 1-point improvement from baseline in superficial, vertical, perioral rhytids based on the 5-point Merz® Scale

SECONDARY OUTCOMES:
Response to Therapy- Subject | Day 0, 7, 14, 30, 60, 90, 120, 150, 180
  Response to therapy on each side of the lip on day 0 (initial treatment), and subsequent post-treatment days 7, 14, 30, 60, 90, 120, 150, 180, as measured by the blinded patient: A 20% improvement from baseline in superficial, vertical, perioral rhytids using a linear analog scale
Severity grading- Evaluator | 6 months
  Severity grading by a blinded evaluator employing standardized photography in combination with the 5-point Merz® Scale
VISIA complexion analysis | Day 0, Day 30
  VISIA complexion analysis (Canfield Imaging Systems, Fairfield, New Jersey) on day 0 (initial treatment), day 30 and when the patient's perioral fine lines have returned to baseline. VISIA analysis will be used to grade the patient's skin by measuring the wrinkles and generating a percentile score.

CONTACTS AND LOCATIONS:
Overall Officials: Corey S. Maas, M.D., Principal Investigator — The Maas Clinic
Locations (1):
- The Maas Clinic, San Francisco, California, United States